CLINICAL TRIAL: NCT00403143
Title: Do Blue-Blocking Lenses Block Colour From Our Lives? A Randomised Controlled Study Measuring Colour Vision Using the Gold Standard Colour Vision Test (an Anomaloscope)in Patients With Blue Light Filtering Intraocular Lenses (Tinted Yellow) and Comparing This With Patients Inserted With Clear, Non Blue Light Filtering Intraocular Lenses During Cataract Surgery
Brief Title: Do Blue-Blocking Lenses Block Blue Colour From Our Lives?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Opa/23
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Blindness
Keywords: intraocular lens, colour vision, blue-light filtering
MeSH Terms: conditions — Blindness | interventions — Cataract Extraction

INTERVENTIONS:
Procedure: cataract surgery

SUMMARY:
To measure colour vision in patients with a blue light filtering lens implant in one eye and non-tinted implant in the other eye (and compared this group with a control group with bilateral non-tinted implants) and to determine whether blue light filtering lenses limit colour vision

DETAILED DESCRIPTION:
As we all age, the natural lens inside our eyes becomes denser, hazy and more yellow in colour. In other words, cataracts develop. In order to enable clear vision again, cataract surgery is performed. This involves removing the natural lens from the eye and replacing it with a synthetic lens implant inside the eye. Cataract surgery with insertion of a lens implant was first done in 1948 but didn't become routine until the early 1980s. Around this time, awareness about the harmful effects of UV light were raised and by 1986, lens implants routinely had a UV filter incorporated into them.1 As early as 1992, a study examining patients who had had a high occupational exposure to blue and visible light, concluded that there is a positive association between long term exposure to visible light and age related wear and tear change at the back of the eye, termed age related macular degeneration (AMD).2 This theory was supported by several studies which have reported an increased rate of progression of AMD in patients after cataract surgery with a clear lens implant (It is known that clear lens implants transmit more blue light to the back of the eye compared with the natural aging lens).3 Laboratory studies in 2000 showed that blue light causes damage to aging retinal cells (the nerve cells at the back of the eye which are important in enabling us to see), more so than green light or white light.4 Experimental studies with rats also showed that exposure to blue light was 30 times more damaging to retinal cells compared with yellow light.5 A further laboratory study in 2004 confirmed that by protecting aging retinal cells with a blue light filtering lens, damage caused by blue light is prevented.6 Yellow tinted, blue light filtering lens implants have been in production since 1991, first by Hoya in Tokyo and now by Alcon as well. Alcon produce the Acrysof Natural lens implant which has been designed to mimic the 53 year old natural lens and which received FDA and CE approval in 2003. To date, over 2 million of these lenses have been implanted in patients world wide.7 Although these lens implants are sometimes used in patients having cataract surgery in the UK, this is not yet routine. One of the concerns about them is whether or not they limit colour vision in any way. There have been some studies examining this and so far, none of them have found a statistically significant difference in the colour vision between patients with non-tinted lens implants and blue-filtering lens implants.8,9,10 However, none of the studies thus far, have employed colour vision testing with an anomaloscope (which is considered to be the gold standard colour vision test).11 In addition, none of them have taken into account the level of capsular opacification (the capsule is a cling film bag-like structure that supports the lens implant inside the eye and can over a period of time, become thickened and hazy following cataract surgery) and the level of macular pigment (yellow pigment which we have on the centre part of the back of our eyes which is thought to contribute towards filtering blue light) in patients' eyes.

Age related macular degeneration is already the commonest cause of blindness in the UK. It is a growing problem, particularly with our aging population and increasing levels of ambient light which we are exposed to in our daily lives. Although the evidence is strongly in favour of filtering blue light and the need for protective measures against AMD are pressing, we need to be satisfied that there are no adverse effects of blocking blue from our lives.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had uncomplicated cataract surgery in one eye and have a cataract in the other eye
* patients who are over 18 years of age
* patients who are fully able to independently give consent to have surgery

Exclusion Criteria:

* patients who have any other ocular co-morbidity that may account for reduction in vision in either eye (as this may confound the condition)
* patients who are colour blind
* patients who suffered previous post-operative complications
* patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
To objectively determine whether colour vision is reduced with a blue-light filtering
intraocular lens compared with a colourless intraocular implant in cataract surgery

SECONDARY OUTCOMES:
To determine whether patients subjectively are able to tell whether they have been
implanted with yellow tinted intraocular lens during their cataract surgery or colourless one

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Vafidis, MA FRCS FRCOphth, Study Director — London North West Healthcare NHS Trust
Locations (1):
- North West London Hospitals NHS Trust, London, United Kingdom